CLINICAL TRIAL: NCT03643965
Title: A Randomized, Double-blind, Placebo Controlled Study to Evaluate Efficacy and Safety of Nefecon in Patients With Primary IgA (Immunoglobulin A) Nephropathy at Risk of Progressing to End-stage Renal Disease (NefIgArd)
Brief Title: Efficacy and Safety of Nefecon in Patients With Primary IgA (Immunoglobulin A) Nephropathy
Acronym: Nefigard
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nef-301
Record Dates: First submitted 2018-08-08; First posted 2018-08-23 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Primary IgA Nephropathy
Keywords: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nefecon (Experimental): Nefecon 16 mg once daily by mouth for 9 months.
  Interventions: Drug: Nefecon
- Placebo oral capsule (Placebo Comparator): Placebo oral capsule once daily by mouth for 9 months.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Nefecon — Nefecon 16 mg for daily administration by mouth for 9 months.
  Other Names: Budesonide modified released capsule
  Arms: Nefecon
Drug: Placebo oral capsule — Placebo capsules for daily administration by mouth for 9 months.
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
The overall aim of the study is to evaluate the efficacy, safety, and tolerability of Nefecon 16 mg per day in the treatment of patients with primary IgAN (Immunoglobulin A nephropathy) at risk of progressing to end-stage renal disease (ESRD), despite maximum tolerated treatment with renin-angiotensin system (RAS) blockade using angiotensin converting enzyme inhibitors (ACEIs) or angiotensin II type I receptor blockers (ARBs).

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy, safety, and tolerability of oral Nefecon compared to matching placebo in patients with primary IgAN on a background of optimized RAS inhibitor therapy. The study will consist of 2 parts, Part A and Part B. Part A will include a 9 month blinded Treatment Period, and a 3-month Follow up Period. Part B of the study will consist of a 12-month observational Follow up Period; no study drug will be administered during Part B. Part A and B will be blinded. Safety will be monitored by an independent Data Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients ≥18 years
2. Biopsy-verified IgA nephropathy
3. Stable dose of RAS inhibitor therapy (ACEIs and/or ARBs) at the maximum allowed dose or Maximum Tolerated Dose (MTD) according to the 2012 KDIGO (Kidney Disease: Improving Global Outcomes) guidelines
4. Urine protein creatinine ratio ≥1 g/24hr
5. eGFR ≥35 mL/min per 1.73 m2 and ≤90 mL/min per 1.73 m2 using the Chronic Kidney Diseae Epidemiology Collaboration (CKD-EPI) formula
6. Willing and able to give informed consent

Exclusion Criteria:

1. Systemic diseases that may cause mesangial IgA deposition.
2. Patients who have undergone a kidney transplant.
3. Patients with acute or chronic infectious disease including hepatitis, tuberculosis, human immunodeficiency virus (HIV), and chronic urinary tract infections.
4. Patients with liver cirrhosis, as assessed by the Investigator.
5. Patients with a diagnosis of type 1 or type 2 diabetes mellitus which is poorly controlled.
6. Patients with history of unstable angina, class III or IV congestive heart failure, and/or clinically significant arrhythmia, as judged by the Investigator;
7. Patients with unacceptable blood pressure control defined as a blood pressure consistently above national guidelines for proteinuric renal disease, as assessed by the Investigator
8. Patients with diagnosed malignancy within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krassimir Mitchev, MD, Study Director — Calliditas AB
Locations (142):
- United States (34):
  - University of Alabama at Birmingham, 1720 2nd Ave South, Birmingham, Alabama
  - Univ of Arizona, 1501 N Campbell Ave, Tucson, Arizona
  - Stanford University Medical Center, 777 Welch Rd, Palo Alto, California
  - Los Angeles Biomedical Research Institute at HUMC, 1124 W. Carson Street, Torrance, California
  - University of Colorado Health Science Center, 1200 East 19th Av., Aurora, Colorado
  - Western Nephrology and Metabolic Bone Disease, PC-Westerminster, 8410 Decatur St., Westminster, Colorado
  - Yale University School of Medicine, 330 Cedar Street, New Haven, Connecticut
  - Washington Nephrology Associates-Washington DC, 730 24th Street NW, Washington D.C., District of Columbia
  - University of Florida-Gainesville, Gainesville, Florida
  - Omega Research Maitland, 7912 Forest City Rd., Orlando, Florida
  - Omega Research Maitland, Orlando, Florida
  - Northwestern University the Feinberg School of Medicine, 633 North St. Clair, Chicago, Illinois
  - Northshore University Health System, 2650 Ridge Av., Evanston, Illinois
  - University of Kentucky Medical Center, 800 Rose St, Pavillion H 3rd floor, Lexington, Kentucky
  - University of Louisville-Nephrology, Louisville, Kentucky
  - Kidney Care and Transplant Services of New England, PC, 354 Birnie Av., Springfield, Massachusetts
  - University of Minnesota, 717 Delaware St. SE, Minneapolis, Minnesota
  - Clinical Research Consultants, LLC, 3930 Washington St, Kansas City, Missouri
  - Queens Hospital Centre, Jamaica, New York
  - Icahn School of Medicine at Mount Sinai-James J. Peters VA Medical Center, One Gustave L. Levy Place, New York, New York
  - Columbia Univ Medical Center, Div of Nephrology, 51 Audubon Av, New York, New York
  - Mountain Kidney & Hypertension Assoc, 10 McDowell St, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Clinical & Translational Research Centre, Chapel Hill, North Carolina
  - Southeastern Nephrology-Whiteville, 800 Jefferson St, Whiteville, North Carolina
  - Southeastern Nephrology Associates-Wilmington, 1302 Medical Center Drive, Wilmington, North Carolina
  - Cleveland Clinic, Glickman Urological & Kidney Institute, 9500 Euclid Av., Cleveland, Ohio
  - The Ohio State University (OSU), Wexner Medical Center, 410 West 10th Av., Columbus, Ohio
  - Oregon Health & Science University, 3181 SW Sam Jackson Park Rd, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, 211 S. 9th Street, Philadelphia, Pennsylvania
  - Allegheny General Hospital, 4800 Friendship Av., Pittsburgh, Pennsylvania
  - Nephrology Associates, P.C., 28 White Bridge Rd, Nashville, Tennessee
  - Renal Disease Research Institute, 1250 Eighth Av. #135, Fort Worth, Texas
  - University of Vermont, Burlington, Vermont
- Argentina (6):
  - Hospital Britanico de Buenos Aires, Pedriel 74, Capital Federal
  - Clinica Priv Velez Sarsfield, Córdoba
  - Hospital Privado-Centro Medico de Cordoba, Naciones Unidas 346, Nefrologia piso 1, Córdoba
  - Sanatorio Allende, Hipolito Yrigoyen 384, 2 Piso, Córdoba
  - Hospital Universitario Austral, Unidad de Investigacion Clinica, Av. J.D. Peron 1500, piso 4, Pilar
  - Clinico de Nefrologia, Urologia Y Enfermedades Cardiovasculares, Av. Gdor Freyre 3074, Santa Fe
- Australia (9):
  - Monash Medical Centre, Clayton, Victoria
  - Royal Adelaide Hospital, Port Rd., Adelaide
  - Box Hill Hospital, Dept of Renal Medicine, Arnold Str 5, Box Hill
  - Austin Health, Dept of Nephrology, 145 Studley Rd., Heidelberg
  - Melbourne Health, Royal Melbourne Hospital, Dept of Nephrology,Grattan Str., Parkville
  - Prince of Wales Hospital, Nephrology Dept, Parkes 3 West, Randwick
  - Western Health, Western Hospital-Sunshine Hospital, 176 Furlong Rd, Level 3, WHCRE Building, St Albans
  - Westmead Hospital, Dept of Renal Medicine, Hawkesbury Rd., Westmead
  - Metro South Hospital and Health Service via Princess Alexandra Hospital, Dept of Nephrology, 199 Ipswich Rd., Woolloongabba
- Belarus (4):
  - Brest Regional Hospital, 7 Meditsinskaya str., Brest
  - Grodno Regional Clinical Hospital, 52 Bulvar Leninskogo Komsomola, Grodno
  - Gomel Regional Clinical Hospital, 5 Brat'ev Lizukovyh str., Homyel
  - 4-th N.E. Savchenko City Clinical Hospital, 110, R. Luxemburg str., Minsk
- Belgium (5):
  - University Hospital Erasmus (Brussels), Recherche Clinique Nephrologie Transplantation, Route de Lennik 808, Brussels
  - Cliniques Universitaires Saint-Luc, Nephrology Dept, Av. Hippocrate 10, Brussels
  - University Hospital Gent, Dept of Medical Nephrology, Corneel Heymanslaan 10, Ghent
  - Centre Hospitalier Universitaire de Liege, Nephrology Dept. Domaine Universitaire de Sart-Tilman, Liège
  - AZ Delta, Wilgenstraat 2, Roeselare
- Canada (10):
  - Royal Inland Hospital, Kidney Clinic, 7 South, 311 Columbia Street, Kamloops, British Columbia
  - Interior Health-Kelowna General Hosp (IH KGH), 2268 Pandosy Str., Kelowna, British Columbia
  - Vancouver Coastal Health Authority, Gordon and Leslie Diamond Health Care Centre, 5 th floor, Diamond Building, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, 1276 South Park St, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Hospital Maisonneuve-Rosemont, CNIB 3rd Floor, 1929 Bayview Avenue, Toronto, Ontario
  - Toronto General Hospital, University Health Network, 200 Elizabeth St, 8 N-849, Toronto, Ontario
  - CISSS de la Monteregie-Centre-Hopital Charles LeMoyne, Room E-304, 3120 Taschereau Blvd, Greenfield Park, Quebec
  - CHUQ-L'Hotel Dieu de Quebec, 11 côte du Palais, Québec, Quebec
  - Centre Hospiitalier Universitaire de Sherbrooke (CHUS), 3001, 12e Avenue Nord, Sherbrooke, Quebec
- Czechia (5):
  - Fakultni nemocnice Brno, Interni gastroenterologicka klinika, Jihlavska 20, Brno
  - Fakultni nemocnice Hradec Kralove, Sokolska 581, Hradec Králové
  - Fakultni nemocnice Olomouc, I.P. Pavlova 185/6, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Linterni klinika, Srobarova 1150/50, Prague
  - Vseobecna fakultni nemocnice v Praze, Klinik nefrologie, U Nemocnice 499/2, Prague
- Finland (3):
  - Helsinki University Central Hospital (HUCH), Nephrology Clinic, Meilahti Triangle Hospital, Helsinki
  - Study Cor Oy, Hoitajantie 4, Jyväskylä
  - Tampere University Hospital, P O Box 2000, Munuaiskeskus, Erakennus, 1. kerros, Tampere
- France (6):
  - Centre Hospitalier Boulogne sur Mer, 4eme etage Batiment Administratif, Allee Jacques Monod, Boulogne-sur-Mer
  - CHU Grenoble-Hopital Michallon, Service Nephrologie-Hemodialyse-Aphereses-Transplantation Renale, Boulevard de la Chantourne CS 10217, Grenoble
  - Lapeyronie Hospital, Univ Hospital Montpellier, 371 Av. du Doyen Gaston Giraud, Montpellier
  - Hopital Bichat-Claude Bernard, Service de Nephrologie, 46 rue Henri Huchard, Paris
  - Chu St Etienne-Hopital Nord, Service de Nephrologie Dialyse Transplantation renale, Av. Albert Raimond, Saint-Priest-en-Jarez
  - Centre Hospitalier de Valenciennes, Service de Nephrologie-Medecine Interne, Av. Desandrouin BP 379, Valenciennes
- Germany (7):
  - Uniklinik RWTH Aachen, Medizinische Klinik II, Pauwelsstrasse 30, Aachen
  - Universitaetsklinikum Carl Gustav Carus Dresden, Medizinische Klinik III, Nephrologie, Fetscherstr. 74, Dresden
  - Universitaetsklinikum Erlangen, Medizinisches Klinik 4, Ulmenweg 18, Erlangen
  - Universitaetsklinikum Heidelberg-Nephrologie, Renal Clinic, Im Neuenheimer Feld 162, Heidelberg
  - Universitatsklinik Schleswig-Holstein-Campus Lubek, Medizinische Klinik I, Nephrologie, Ratzeburger Allee 160, Lübeck
  - University Clinic Munich, LMU-Inner City Medical Polyclinic, Nephrologisches Zentrum, Medizinische Klinik und Poliklinik IV, Munich
  - Universitaetsklinikum Regensburg, Abteilung für Nephrologie, Franz-Josef-Strauss Allee 11, Regensburg
- Greece (7):
  - General Hospital of Athens-Laiko, Nephrology Clinic, 17 Agiou Thoma Street, Athens
  - University Hospital of Heraklion, Nephrology Clinic, Diastaurosi Staurakion-Vouton, Heraklion
  - University General Hospital of Ioannina, Nephrology Clinic, Leof. Stavros Niarchou, Ioannina
  - University Hospital of Larissa Medical School, Nefrology Clinic, Mezourlo, Larissa
  - General Hospital of Nikaia Ag. Panteleimon, Nephrology Clinic, Mantouvalou 3 Str., Nikaia
  - University General Hospital of Patras, Rio, Pátrai
  - Hippokration General Hosp of Thessaloniki, Nephrology Clinic, 49 Konstantinoupoleos Str, Thessaloniki
- Italy (4):
  - Azienda Ospedale Policlinico di Bari, Bari
  - ASST di Lecco, Presidio Ospedaliero Alessandro Manzoni, Via dell´Eremo 9/11, Lecco
  - Ospedale San Carlo Borromeo, Via Pio II, 3, Milan
  - Istituti Clinici Scientifici Maugeri Spa-Societa Benefit, Div. di Nephrologia ed Emodialist, Via S. Maugeri 10, Pavia
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne-Szpital Gdanskiego Uniwersytetu Medycznego, Gdansk
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Centralny Szpital Kliniczny, Uniwersytetu Medycznego w Lodzi, ul Pomorska 251, Lodz
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Oddzial Kliniczny Nefrologiczny, Hipertensjologii i Chorob Wewnetrznych, ul. Zolnierska 18, Olsztyn
  - Sonomed Sp. z.o.o. ul. Bandurskiego 98/U12, Szczecin
- South Korea (7):
  - Dong-A University Hospital, Won Suk An, 26 Daesingongwon-Ro Seogu, Busan
  - Kyungpook National University Hospital, 130 Dongdeok-ro Jung-gu, Daegu
  - Chungnam National University Hospital, 282 Munhwa-ro, Jung-gu, Daejeon
  - Hallym University Sacred Heart Hospital,22 Gwanpyeong-ro 170 beon-gil, Dongan-gu, Anyang-si, Gyeonggi-do
  - Seoul National University Hospital, 101 Daehak-Ro, Jongno-Gu, Seoul
  - Seoul St. Mary´s Hospital, 222 Banpo-Daero, Seocho-gu, Seoul
  - Chung-Ang University Hospial, 102 Heukseok-ro, Dongiak-gu, Seoul
- Spain (7):
  - Hospital Universitario Fundacion Alcorcon, C/Budapest 1, Alcorcón
  - Hospital del Mar, Passeig Maritim 25-29, Barcelona
  - Hospital Universitario Vall d´Hebron, Passeig Vall d´Hebron 119-129, Barcelona
  - Hospital Clinic Barcelona, Escalera 12, Planta 5, Calle Villaroel 170, Barcelona
  - Hospital Universitari Arnau de Vilanova, Avenida Alcalde Rovire Roure 80, Lleida
  - Hospital General Universitario Gregorio Maranon, Servicio de Nefrologica, C/Dr. Esquerdo 46, Madrid
  - Hospital 12 de Octubre, Residencia General (Sotano 1)-Area de Ensayos Clinicos, Avda. Cordoba s/n, Madrid
- Sweden (5):
  - Sahlgrenska University Hospital, Njurmottagningen, Vita Stråket 12, Gothenburg
  - Universitetssjukhuset Linköping, Njurmedicinska kliniken, Linköping
  - Karolinska University Hospital-Huddinge, Njur-KBC M87, Stockholm
  - Danderyds sjukhus, Njurmedicinska kliniken, Stockholm
  - Uppsala University Hospital, Dept of Nephrology, ing 30, plan 5, Uppsala
- Taiwan (4):
  - Kaohsiung Medical Univ Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, No 2 Yude Rd, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, No 138 Sheng Li Rd, Tainan
- Turkey (Türkiye) (5):
  - Cukurova University Medical Faculty, Dept of Internal Disease, Div of Nephrology, Balcali, Adana
  - Istanbul University Cerrahpasa, Medical Faculty-Dept of Internal Disease, Fatih-Cerrahpasa, Kocamustafapasa Caddesi No 53, Istanbul
  - Ege University Med Faculty Dept of Internal Disease, Div of Nephrology, Izmir
  - Erciyes University Faculty of Medicine,Semiha Kibar Organ Nakli ve Dyaliz Hastanesi, Kosk Mah. prof dr Turhan Feyziogly Cad. no 42, Kayseri
  - Kocaeli University Medical School-Internal Medicine, Nephrology, Umuttepe Yerleskesi, Kocaeli
- United Kingdom (10):
  - Belfast City Hospital, 51 Lisburn Rd, Belfast
  - Southmead Hospital, Southmead Rd, Westbury-on-Trym, Bristol
  - Queen Elizabeth University Hosp-Glasgow, Glasgow Clin Research Facility 5th floor, Institute of Neurosciences, Glasgow
  - Gloucestershire Royal Hospital, Great Western Rd, Gloucester
  - St James´s University Hospital, Beckett St., Leeds
  - Leicester General Hospital, John Walls Renal Unit, Gwendolen Rd, Leicester
  - The Royal London Hospital, Whitechapel, London
  - University of Manchester, Manchester Royal Infirmary, Oxford Rd, Manchester
  - Nottingham City Hospital, Hucknall Rd, Nottingham
  - Northern General Hospital, Herries Rd., Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fellstrom BC, Barratt J, Cook H, Coppo R, Feehally J, de Fijter JW, Floege J, Hetzel G, Jardine AG, Locatelli F, Maes BD, Mercer A, Ortiz F, Praga M, Sorensen SS, Tesar V, Del Vecchio L; NEFIGAN Trial Investigators. Targeted-release budesonide versus placebo in patients with IgA nephropathy (NEFIGAN): a double-blind, randomised, placebo-controlled phase 2b trial. Lancet. 2017 May 27;389(10084):2117-2127. doi: 10.1016/S0140-6736(17)30550-0. Epub 2017 Mar 28. PMID 28363480
- [Derived] Zhang H, Lafayette R, Wang B, Ying L, Zhu Z, Stone A, Kristensen J, Barratt J. Efficacy and Safety of Nefecon in Patients with IgA Nephropathy from Mainland China: 2-Year NefIgArd Trial Results. Kidney360. 2024 Dec 1;5(12):1881-1892. doi: 10.34067/KID.0000000583. Epub 2024 Oct 9. PMID 39724565
- [Derived] Lafayette R, Kristensen J, Stone A, Floege J, Tesar V, Trimarchi H, Zhang H, Eren N, Paliege A, Reich HN, Rovin BH, Barratt J; NefIgArd trial investigators. Efficacy and safety of a targeted-release formulation of budesonide in patients with primary IgA nephropathy (NefIgArd): 2-year results from a randomised phase 3 trial. Lancet. 2023 Sep 9;402(10405):859-870. doi: 10.1016/S0140-6736(23)01554-4. Epub 2023 Aug 14. PMID 37591292
- [Derived] Liao J, Zhou Y, Xu X, Huang K, Chen P, Wu Y, Jin B, Hu Q, Chen G, Zhao S. Current knowledge of targeted-release budesonide in immunoglobulin A nephropathy: A comprehensive review. Front Immunol. 2023 Jan 4;13:926517. doi: 10.3389/fimmu.2022.926517. eCollection 2022. PMID 36685528
- [Derived] Barratt J, Lafayette R, Kristensen J, Stone A, Cattran D, Floege J, Tesar V, Trimarchi H, Zhang H, Eren N, Paliege A, Rovin BH; NefIgArd Trial Investigators. Results from part A of the multi-center, double-blind, randomized, placebo-controlled NefIgArd trial, which evaluated targeted-release formulation of budesonide for the treatment of primary immunoglobulin A nephropathy. Kidney Int. 2023 Feb;103(2):391-402. doi: 10.1016/j.kint.2022.09.017. Epub 2022 Oct 19. PMID 36270561

RESULTS

PARTICIPANT FLOW:
Period: Part A
Arm/Group | Nefecon | Placebo Oral Capsule
Started | 182 | 182
Completed | 175 | 174
Not Completed | 7 | 8
Period: Part B
Arm/Group | Nefecon | Placebo Oral Capsule
Started | 175 | 174
Completed | 161 | 165
Not Completed | 14 | 9

BASELINE CHARACTERISTICS:
Population: Full analysis set - Global study
Groups:
- Total: Total of all reporting groups
Arm/Group | Nefecon | Placebo Oral Capsule | Total
Number analyzed (Participants) | 182 | 182 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (10.78) | 41.6 (10.65) | 42.7 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 59 | 124
  Male | 117 | 123 | 240
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 43 | 40 | 83
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 138 | 137 | 275
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Baseline Urine protein to creatinine ratio (UPCR) [Geometric Mean (Inter-Quartile Range); unit: g/gram] | 1.300 [0.902 to 1.764] | 1.264 [0.877 to 1.737] | 1.282 [0.892 to 1.752]
Baseline Estimated glomerular filtration rate (eGFR) [Geometric Mean (Inter-Quartile Range); unit: ml/min/1.73 m2] | 56.006 [45.497 to 70.972] | 55.565 [45.957 to 67.735] | 55.785 [45.929 to 69.839]

OUTCOME MEASURES:

1. Primary Outcome: Part A: Ratio of Urine Protein to Creatinine Ratio (UPCR) at 9 Months Compared to Baseline
Description: Part A primary endpoint: The ratio of Urine Protein to Creatinine Ratio (UPCR) (based on 24-hour urine collections) at 9 months following the first dose of study drug compared to baseline.
  Ratio being: UPCR at 9 months in g/gram divided with UPCR at Baseline in g/gram
Time Frame: 9 months
Population: Full analysis set - global study - Part A
Measure: Geometric Least Squares Mean (96% Confidence Interval); unit: ratio
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 97 | 102
ratio | 0.69 [0.61 to 0.79] | 0.95 [0.83 to 1.08]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Ratio of UPCR at 9 months compared to baseline for Nefecon compared to Placebo; p = 0.0003, MMRM model; Ratio of geometric LS means = 0.73, 96% CI 2-sided [0.61 to 0.88]

2. Primary Outcome: Part B: Time-weighted Average of Estimated Glomerular Filtration Rate (eGFR)
Description: Part B Primary endpoint: Time-weighted average of estimated glomerular filtration rate (eGFR) recordings observed at each time point over 2 years. The eGFR (CKD-EPI) at 2 years (which must have been repeated to provide a second value obtained within 14 to 35 days) was the geometric mean of the 2 assessments.
Time Frame: Up to 2 years and 1 month
Population: Full analysis set - global study - Part B
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 182 | 182
mL/min/1.73m2 | 0.96 [0.93 to 0.98] | 0.87 [0.84 to 0.89]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Time-weighted average of eGFR, Nefecon compared to Placebo; p < 0.0001, robust regression; Ratio of geometric LS means = 1.10, 95% CI 2-sided [1.06 to 1.15]

3. Secondary Outcome: Part A: Ratio of eGFR at 9 Months
Description: Part A: Ratio of eGFR at 9 months compared to baseline calculated using the CKD-EPI formula.
Time Frame: 9 months
Population: Full analysis set - global study - Part A
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 97 | 102
mL/min/1.73m2 | 1.00 [0.96 to 1.03] | 0.93 [0.90 to 0.96]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Ratio of eGFR at 9 months comparison of Nefecon to Placebo; p = 0.0014, robust regression; Ratio of geometric LS means = 1.07, 95% CI 2-sided [1.03 to 1.13]

4. Secondary Outcome: Part A: Ratio of eGFR at 12 Months
Description: Part A: Ratio of eGFR at 12 months compared to baseline calculated using the CKD-EPI formula.
Time Frame: 12 months
Population: Full analysis set - global study - Part A
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 97 | 102
mL/min/1.73m2 | 0.97 [0.93 to 1.01] | 0.91 [0.88 to 0.95]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Ratio of eGFR at 12 months comparison of Nefecon to Placebo; p = 0.0106, robust regression; Ratio of geometric LS means = 1.07, 95% CI 2-sided [1.01 to 1.13]

5. Secondary Outcome: Part A: Ratio of Urine Albumin to Creatinine Ratio (UACR) at 9 Months
Description: Part A: Ratio of urine albumin to creatinine ratio (UACR) at 9 months compared to baseline.
Time Frame: 9 months
Population: Full analysis set - global study - Part A
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: g/gram
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 97 | 102
g/gram | 0.64 [0.55 to 0.75] | 0.93 [0.80 to 1.09]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Ratio of UACR at 9 months comparison of Nefecon to Placebo; p = 0.0005, MMRM model; Ratio of geometric LS means = 0.69, 95% CI 2-sided [0.55 to 0.86]

6. Secondary Outcome: Part B: Time to 30% Reduction in eGFR
Description: Part B: Time to 30% reduction from baseline in eGFR (CKD-EPI) confirmed by a second value.
  For clarity: Please note that the number of patients with a 30% reduction is presented with statistical analysis of the time to 30% reduction.
Time Frame: Over 2 years
Population: Full analysis set - global study - Part B
Measure: Number; unit: Participants
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 182 | 182
Participants | 21 | 39
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Time to 30% reduction in eGFR comparison Nefecon to Placebo; p = 0.0028, Cox proportional hazards model; Cox proportional hazards model with individual patient censoring weighting; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.26 to 0.75]

7. Secondary Outcome: Part B: Time to Receiving Rescue Medication.
Description: Part B: Time from the first dose of study drug until receiving rescue medication.
  For clarity: Please note that the number of patients receiving rescue medication is presented with statistical analysis of the time to receiving rescue medication.
Time Frame: Over 2 years
Population: Full analysis set - global study - Part B
Measure: Number; unit: Participants
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 182 | 182
Participants | 15 | 20
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Time to receiving rescue medication comparison Nefecon to Placebo; p = 0.2647, Cox proportional hazards model; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.34 to 1.33]

8. Secondary Outcome: Part B: Ratio of UPCR Compared to Baseline Averaged Over Time Points Between 12 and 24 Months
Description: Part B: Ratio of UPCR, UACR, and eGFR (CKD-EPI) compared to baseline averaged over time points between 12 and 24 months, inclusive, following the first dose of study drug
Time Frame: 12, 18 and 24 months
Population: Full analysis set - global study - Part B
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: g/gram
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 172 | 173
g/gram | 0.60 [0.54 to 0.66] | 1.01 [0.91 to 1.12]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Ratio of UPCR compared to baseline averaged over time points between 12 and 24 months, comparison Nefecon vs Placebo; p < 0.0001, MMRM model; Ratio of geometric LS means = 0.59, 95% CI 2-sided [0.51 to 0.68]

9. Secondary Outcome: Part B: Ratio of UACR Compared to Baseline Averaged Over Time Points Between 12 and 24 Months
Description: as for outcome 8
Time Frame: 12 to 24 months
Population: Full analysis set - global study - Part B
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: g/gram
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 172 | 173
g/gram | 0.52 [0.46 to 0.58] | 0.96 [0.86 to 1.08]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Ratio of UACR compared to baseline averaged over time points between 12 and 24 months, Nefecon vs Placebo; p < 0.0001, MMRM model; Ratio of geometric LS means = 0.54, 95% CI 2-sided [0.45 to 0.63]

10. Secondary Outcome: Part B: Ratio of eGFR Compared to Baseline Averaged Over Time Points Between 12 and 24 Months
Description: Part B: Ratio of UPCR, UACR, and eGFR (CKD-EPI) compared to baseline averaged over time points between 12 and 24 months, inclusive, following the first dose of study drug;
Time Frame: 12 to 24 months
Population: Full analysis set - global study - Part B
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: mL/min/1.73m2
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 163 | 166
mL/min/1.73m2 | 0.93 [0.90 to 0.96] | 0.84 [0.81 to 0.86]
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Ratio of eGFR compared to baseline averaged over time points between 12 and 24 months, comparison Nefecon vs Placebo; p < 0.0001, robust regression; Ratio of geometric LS means = 1.11, 95% CI 2-sided [1.06 to 1.16]

11. Secondary Outcome: Part B: Proportion of Patients Without Microhematuria
Description: Part B: Proportion of patients without microhematuria in at least 2 of the following time points: 12, 18, and 24 months following the first dose of study drug
Time Frame: 12 to 24 months
Population: Full analysis set - global study - Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 182 | 182
Participants | 94 | 59
Statistical Analysis 1: Comparison: Nefecon vs Placebo Oral Capsule; Test type: Other — Proportion of patients without microhematuria, comparison Nefecon vs Placebo; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.6 to 4.1]

12. Secondary Outcome: Part B: Short Form 36 (SF-36) Quality of Life Assessment at 9 Months.
Description: Part B: Short Form 36 (SF-36) quality of life assessment at 9 and 24 months.
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used. It consists of eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions.
  Higher scores indicate better health. Scores represent the percentage of total possible score achieved.
Time Frame: 9 months
Population: Full analysis set - global study - Part B
Measure: Mean (Standard Deviation); unit: Percentage of total possible score
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 170 | 170
Percentage of total possible score
  Bodily Pain | 54.353 (9.0306) | 54.659 (9.2387)
  General Health | 47.058 (9.6373) | 48.014 (10.0120)
  Mental Component Summary | 49.564 (9.2834) | 49.760 (8.8974)
  Mental Health | 50.226 (8.9539) | 50.099 (8.8483)
  Physical Component Summary | 52.257 (7.2188) | 53.732 (6.5876)
  Physical Functioning | 52.722 (6.7370) | 54.276 (5.2243)
  Role Emotional | 49.574 (9.4322) | 50.393 (8.3001)
  Role Physical | 51.028 (8.0207) | 52.693 (6.6600)
  Social Function | 50.941 (8.3606) | 51.707 (7.9259)
  Vitality | 51.826 (10.0909) | 53.490 (9.3987)

13. Secondary Outcome: Part B: Short Form 36 (SF-36) Quality of Life Assessment at 24 Months.
Description: as for outcome 12
Time Frame: 24 months
Population: Full analysis set - global study - Part B
Measure: Mean (Standard Deviation); unit: Percentage of total possible score
Arm/Group | Nefecon | Placebo Oral Capsule
Number analyzed (Participants) | 159 | 164
Percentage of total possible score
  Bodily Pain | 53.385 (9.6352) | 53.208 (9.9811)
  General Health | 47.038 (9.3450) | 47.214 (9.9564)
  Mental Component Summary | 51.246 (8.1362) | 49.743 (10.2184)
  Mental Health | 51.691 (8.2104) | 50.294 (10.0007)
  Physical Component Summary | 51.443 (7.5200) | 51.993 (7.1783)
  Physical Functioning | 52.665 (7.6364) | 53.059 (6.9006)
  Role Emotional | 50.322 (8.4690) | 49.333 (10.0789)
  Role Physical | 50.948 (7.8921) | 50.722 (8.8255)
  Social Function | 51.949 (7.9677) | 51.471 (8.9304)
  Vitality | 53.291 (8.8558) | 52.364 (10.0023)

ADVERSE EVENTS:
Time Frame: AEs were recorded from time of first dose of study treatment until 2 years after first dose (end of study). Treatment emergent AEs were those that occurred after the first dose of study drug until 14 days after the last dose, including tapering. SAEs were recorded from time of patient informed consent until end of study, i.e until 2 years and 3 months (including follow-up period)
Description: Treatment emergent SAEs are listed on Clinicaltrial.gov.
Arm/Group | Nefecon | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 1/182 | 0/182
Serious Adverse Events (participants affected / at risk) | 18/182 | 9/182
Other Adverse Events (participants affected / at risk) | 108/182 | 69/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nefecon (N=182) | Placebo Oral Capsule (N=182)
Corona virus infection (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Campylobacter colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nefecon (N=182) | Placebo Oral Capsule (N=182)
Edema peripheral (General disorders) | 28 | 7
Hypertension (Vascular disorders) | 21 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 | 7
Acne (Skin and subcutaneous tissue disorders) | 20 | 2
Nasopharyngitis (Infections and infestations) | 17 | 19
Headache (General disorders) | 19 | 14
Upper respiratory tract infection (Infections and infestations) | 10 | 10
Dyspepsia (Gastrointestinal disorders) | 13 | 4
Weight increased (General disorders) | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4
Insomnia (Psychiatric disorders) | 10 | 7
Fatigue (General disorders) | 10 | 7
Diarrhea (Gastrointestinal disorders) | 9 | 10
Rash (Skin and subcutaneous tissue disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03643965/Prot_SAP_000.pdf